CLINICAL TRIAL: NCT04596306
Title: Laparoscopic Cholecystectomy for Acute Calculous Cholecystitis in the Elderly: More Complex But Equally Safe and Effective. A Retrospective Study on 879 Patients.
Brief Title: Laparoscopic Cholecystectomy for Acute Calculous Cholecystitis in the Elderly: A Retrospective Study.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Dario Tartaglia, Ph.D.; M.D., Researcher and Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: DT- 02- 2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UNDER 70 Y-O
  Interventions: Procedure: Laparoscopic Cholecystectomy
- OVER 70 Y-O
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Laparoscopic Cholecystectomy

SUMMARY:
With the progressive aging of the population in industrialized countries, acute calculous cholecystitis (ACC) has been constantly increasing among elderly. Because ACC is the most common complication of biliary gallstone disease and the population will become older, ACC in elderly is expected to increase. In 2017, the incidence of gallstone disease in Italian population is was 18.8% in women and 9.5% in men; the prevalence was 15% and 24% at 70 years and 24% and 35% at 90 years for males and females respectively. Since the increase in age is often associated with an increase in comorbidity, fragility, surgery related complications, morbidity and mortality, the surgical indication for gallstone is still debated and often based on anesthetic risk. In order to avoid surgery for elderly and high-risk patients, alternative treatments to surgery have been developed. The present study aimed to compare two groups of patients with acute calculous cholecystitis undergone laparoscopic cholecystectomy, under and over 70 years old and to assess whether laparoscopy can offer the same safety and efficacy to older people.

ELIGIBILITY:
Inclusion Criteria:

* acute calculous cholecystitis

Exclusion Criteria:

* tumors of the biliary tract

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic cholecystectomy for acute calculous cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
In-hospital morbidity | 30 day
In-hospital mortality | 30 day

SECONDARY OUTCOMES:
conversion to open rate | 30-day
length of stay | 30-day
major complication rate | 30-day

CONTACTS AND LOCATIONS:
Locations (1):
- AOUPisana, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided